CLINICAL TRIAL: NCT03879642
Title: Reducing Hypoglycemia Fear in Parents of Young Kids Via Video-based Telemedicine
Brief Title: Reducing Hypoglycemia Fear in Parents of Young Children With Type 1 Diabetes
Acronym: REDCHiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HD081502 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-03-19 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Parents

STUDY DESIGN:
Intervention Model Description: randomized control pilot using a waitlist control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REDCHiP (Experimental): 10 week video-based telemedicine intervention to reduce parents hypoglycemia fear
  Interventions: Behavioral: REDCHiP
- Waitlist (No Intervention): 10 week no intervention to provide waitlist control condition

INTERVENTIONS:
Behavioral: REDCHiP — 10 week video-based telemedicine intervention to reduce hypoglycemia fear
  Arms: REDCHiP

SUMMARY:
Pilot of a novel video-based telemedicine intervention to reduce fear of hypoglycemia in parents of young children with type 1 diabetes.

DETAILED DESCRIPTION:
This was a two group randomized controlled study using a wait-list control design. All participating parents had the opportunity to receive 10 video-based telemedicine sessions administered over 13 weeks. Study assessments took place at baseline, post-treatment, and 3 month followup. Study outcomes included parent reported hypoglycemia fear, parenting stress, diabetes distress, and child glycated hemoglobin.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children, between 1-6 years old, with type 1 diabetes for at least 6 months, on either multiple daily injections or an insulin pump, and parents speak English

Exclusion Criteria:

* Families of children who are older than 6 years-old and or do not have type 1 diabetes; children follow a conventional insulin regimen

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patton SR, Monzon AD, Noser AE, Clements MA. Physical Activity, Glycemic Variability, and Parental Hypoglycemia Fear in Preschoolers With Type 1 Diabetes. Pediatr Exerc Sci. 2022 Jan 19;34(3):135-140. doi: 10.1123/pes.2021-0046. Print 2022 Aug 1. PMID 35045389
- [Derived] Patton SR, Clements MA, Marker AM, Nelson EL. Intervention to reduce hypoglycemia fear in parents of young kids using video-based telehealth (REDCHiP). Pediatr Diabetes. 2020 Feb;21(1):112-119. doi: 10.1111/pedi.12934. Epub 2019 Nov 3. PMID 31610073
- [Derived] Marker AM, Monzon AD, Nelson EL, Clements MA, Patton SR. An Intervention to Reduce Hypoglycemia Fear in Parents of Young Kids with Type 1 Diabetes Through Video-Based Telemedicine (REDCHiP): Trial Design, Feasibility, and Acceptability. Diabetes Technol Ther. 2020 Jan;22(1):25-33. doi: 10.1089/dia.2019.0244. Epub 2019 Nov 13. PMID 31517512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment in clinic and by telephone
Pre-assignment Details: the study over-recruited the original study protocol by 3 parents; pre-assignment, parents completed baseline assessment measures;
Period: Overall Study
Arm/Group | REDCHiP | Waitlist
Started | 22 | 21
Completed | 19 | 18
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REDCHiP | Waitlist | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: one parent from each condition did not complete all the baseline assessment measures
  years
    number analyzed (Participants) | 21 | 20 | 41
    (all) | 33.81 (4.59) | 36.75 (5.02) | 36.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: one parent from each condition did not complete all baseline assessments
  Participants
    number analyzed (Participants) | 21 | 20 | 41
    Female | 21 | 19 | 40
    Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: one parent in the waitlist control group did not complete this survey
  Participants
    number analyzed (Participants) | 22 | 20 | 42
    Hispanic or Latino | 1 | 1 | 2
    Not Hispanic or Latino | 21 | 17 | 38
    Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 21 | 19 | 40
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia Fear Survey
Description: Hypoglycemia Fear Survey-Parents of Young Children. This is a measure of parents' perceived hypoglycemia fear. Higher scores suggest greater fear (worse outcome). Total possible range: 26-130.
Time Frame: absolute value at post-treatment (week 14)
Population: 43 parents enrolled and were randomized; 36 parents completed the treatment. Therefore number analyzed reflects 36 parents who completed treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | REDCHiP | Waitlist
Number analyzed (Participants) | 18 | 18
units on a scale | 75.94 (18.46) | 70.78 (14.93)
Statistical Analysis 1: Comparison: REDCHiP vs Waitlist; Test type: Superiority; ANOVA; partial eta squared = .117

2. Secondary Outcome: Child Hemoglobin A1c
Description: Child hemoglobin A1c- biological marker of glycemic control
Time Frame: absolute value at post-treatment (week 14)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin cells
Arm/Group | REDCHiP | Waitlist
Number analyzed (Participants) | 18 | 18
percentage of glycated hemoglobin cells | 8.07 (1.30) | 7.97 (0.80)
Statistical Analysis 1: Comparison: REDCHiP vs Waitlist; Test type: Superiority; repeated measures ANOVA; partial eta squared = .005

ADVERSE EVENTS:
Time Frame: through study completion, average 7 months
Description: Adverse event = episodes of prolong low blood glucose value (>1 hour); increase in frequency of any low blood glucose events (glucose <70 mg/dl)
Arm/Group | REDCHiP | Waitlist
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03879642/Prot_SAP_001.pdf